CLINICAL TRIAL: NCT05898373
Title: Phase II, Multi-arm, Open Clinical Study of Recombinant Humanized Anti-HER2 Monoclonal Antibody-MMAE Coupling Agent Vedicitumomab Alone or in Combination for the Treatment of Locally Advanced or Metastatic Salivary Gland Ductal Carcinoma
Brief Title: Vedicitumomab Alone or in Combination for the Treatment of Locally Advanced or Metastatic SDC
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Peking Union Medical College (Other)
Responsible Party: Principal Investigator, Fei Ma, Department of Internal Medicine, Cancer Hospital, Chinese Academy of Medical Sciences, Peking Union Medical College
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: NCC4001; NCC4001 (Other: Ethics Committee of Cancer Hospital)
Record Dates: First submitted 2023-05-15; First posted 2023-06-12 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Salivary Gland Cancer
MeSH Terms: conditions — Salivary Gland Neoplasms | interventions — RC48 antibody

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- vedicitumomab (Experimental): RC48 (2.5 mg/kg every two weeks) intravenously for 6-8 cycles
  Interventions: Drug: vedicitumomab (Edisil, RC48）
- vedicitumomab in combination with pyrrolizidine (Experimental): RC48 （2 mg/kg every two weeks) intravenously for 6-8 cycles in combination with oral HER2 TKI (pyrrolizidine 400 mg qd po)
  Interventions: Drug: vedicitumomab in combination with pyrrolizidine
- RC48 in combination with a platinum-based chemotherapeutic agent (Experimental): RC48 (2 mg/kg every two weeks) in combination with a platinum-based chemotherapeutic agent of the physician's choice (carboplatin 200-250 mg/m2 every two weeks or cisplatin 50 mg/m2 every two weeks) administered intravenously for 6-8 cycles
  Interventions: Drug: RC48 in combination with a platinum-based chemotherapeutic agent
- RC48 in combination with teraplizumab (Experimental): RC48(2 mg/kg every two weeks) in combination with an immune checkpoint inhibitor (teraplizumab, 3 mg/kg every two weeks)
  Interventions: Drug: RC48 in combination with teraplizumab

INTERVENTIONS:
Drug: vedicitumomab (Edisil, RC48） — intravenously for 6-8 cycles before surgery and postoperative radiotherapy, followed by Treatment with injectable recombinant humanized anti-HER2 monoclonal antibody-MMAE coupling agent vedicitumomab (Edisil, RC48) until 1 year or disease progression or intolerable toxicity in locally advanced patients , and until disease progression or intolerable toxicity in metastatic patients .
  Arms: vedicitumomab
Drug: vedicitumomab in combination with pyrrolizidine — vedicitumomab in combination with pyrrolizidine
  Arms: vedicitumomab in combination with pyrrolizidine
Drug: RC48 in combination with a platinum-based chemotherapeutic agent — RC48 in combination with a platinum-based chemotherapeutic agent
  Arms: RC48 in combination with a platinum-based chemotherapeutic agent
Drug: RC48 in combination with teraplizumab — RC48 in combination with teraplizumab
  Arms: RC48 in combination with teraplizumab

SUMMARY:
(1) To apply Bayesian statistics to screen for the most effective treatment regimen containing recombinant humanized anti-HER2 monoclonal antibody-MMAE coupling agent vedicitumomab (Edisil, RC48) for locally advanced or metastatic salivary gland ductal carcinoma expressing HER2 in the near future. (2) To explore biomarkers relevant to the efficacy of recombinant humanized anti-HER2 monoclonal antibody-MMAE-coupled vedicitumomab (Edisil, RC48) in the treatment of HER2-expressing locally advanced or metastatic salivary gland ductal carcinoma.

DETAILED DESCRIPTION:
Using a Bayesian adaptation method based on posterior probabilities, patients will be randomized into four cohorts as follows:

(i) Cohort 1 (RC48 monotherapy group, control group): vedicitumomab monotherapy (2.5 mg/kg, intravenous, Q2w); (ii) Cohort 2 (RC48 + pyrrolitinib group): vedicitumomab (Edexcel, RC48) (2 mg/kg, sedation, Q2w) combined with an oral HER2 TKI (pyrrolitinib 400 mg po qd ); (iii) Cohort 3 (RC48 + platinum group): vedicitumomab (2mg/kg, IV, Q2w) in combination with a physician's choice of platinum-based chemotherapy (carboplatin 200-250mg/m2, IV, Q2w or cisplatin 50mg/m2, IV, Q2w); (iv) Cohort 4 (RC48 + Tremelimumab group): vedicitumomab (2mg/kg, IV, Q2w) in combination with the immune checkpoint inhibitor tremelimumab (3mg/kg, IV, Q2w);

In this study, we will detect HER2 immunohistochemistry, HER2FISH (HER2/CEP17), androgen receptor AR, value-added index ki67, human epidermal growth factor EGFR, basal cytokeratin CK5/6, immune checkpoint PD-L1, type 4 mucin MUC4, recombinant human RAS-related protein, etc. in pre-treatment specimens using traditional immunohistochemistry methods. 5ARAB5A, tumor infiltrating lymphocytes TILs, regulatory T cells Treg and other immune cells, circulating tumor cell DNA (ctDNA) by NGS, blood count, lymphocyte subsets, and HER2 ECD by ELISA. Patients with locally advanced disease were divided into pCR group (complete remission group) and non-pCR group (non-complete remission group) according to their clinical response to treatment, and patients with advanced metastatic disease were divided into PD group (disease progression group) and non-PD group (non-progression group), comparing the differences between the pCR and non-pCR groups, and the differences between the PD and non-PD groups, and exploring the differences with vedicizumab (Edisil, RC48) in monotherapy or combination for salivary gland ductal carcinoma.

ELIGIBILITY:
Inclusion Criteria:

(1) Patients with advanced metastatic salivary gland ductal carcinoma diagnosed histopathologically at the primary site or metastasis; (2) Original paraffin-embedded tumor tissue stained for HER2 at diagnosis, either HER2 1+/HER2 2+/HER2 3+, previous test results (confirmed by the investigator) or test results from the study center are acceptable; (3) ECOG physical status 0 or 1 within 3 days prior to the first dose of study treatment; (4) 18 years of age or older - upper limit; (5) Life expectancy greater than 3 months according to RECIST 1.1 criteria; (6) At least one measurable lesion; and (7) a score of 0 or 1 for ECOG physical status within 3 days prior to the first dose of study treatment. status 0 or 1 within 3 days prior to the first dose of study treatment; ④ 18 years of age or older - no upper limit; ⑤ life expectancy greater than 3 months; ⑥ at least one measurable lesion according to RECIST 1.1 criteria;(7) Female subjects should be surgically sterilized, post-menopausal, or agree to use at least one medically approved contraceptive (e.g., IUD, pill, or condom) during and for 6 months after the study treatment period, and must have a negative blood pregnancy test within 7 days prior to study entry and must be non-lactating. Male subjects should agree to use at least one medically approved contraceptive measure during the study treatment period and for 6 months after the end of the study treatment period; ⑧ Patients must have adequate liver, kidney, bone marrow, heart and lung organ function: bone marrow function: (1) hemoglobin ≥ 90 g/L; (2) absolute neutrophil count ≥ 1.5 × 109/L; (3) platelets ≥ 100 × 109/L Liver function (based on the normal value of the clinical trial center): (1) without liver metastases, serum total bilirubin ≤ 1.5 times ULN; with liver metastases, serum total bilirubin ≤ 3 times ULN (2) without liver metastases, ALT and AST are ≤ 3 times ULN, with liver metastases, ALT and AST are ≤ 5 times ULN Kidney function (based on the normal value of the clinical trial center): (1) blood creatinine ≤ 1.5 times ULN, or 1.5 times ULN, or Cockcroft-Gault formula calculated creatinine clearance (CrCl) ≥ 60 mL/min, or measured 24-hour urine CrCl ≥ 60 mL/min; cardiac function: (1) New York Heart Association (NYHA) classification <3 (2) left ventricular ejection fraction ≥ 50%

Exclusion Criteria:

(i) treatment with an investigational drug or other antibody-coupled drug targeting HER2 at the start of the study drug; (ii) major surgery within 4 weeks prior to the start of the study drug and incomplete recovery; (iii) live vaccination within 4 weeks prior to the start of the study drug or any vaccine planned during the study period (except novel coronavirus vaccine);(iv) an arterial/venous thrombotic event such as cerebrovascular accident (including temporary ischemic attack), deep vein thrombosis, or pulmonary embolism within 6 months prior to study drug administration; (v) major cardiovascular disease (NYHA class 3 or 4 heart failure, second degree or greater heart block, myocardial infarction within the past 12 months, unstable arrhythmia or unstable angina, cerebral infarction within 6 months, etc.); (vi) ongoing unstable controlled systemic disease, including diabetes, hypertension, pulmonary fibrosis, acute lung disease, interstitial lung disease, cirrhosis, etc;(7) Active infection requiring systemic therapy; (8) History of active tuberculosis; (9) Positive human immunodeficiency virus (HIV) test result; (10) Positive hepatitis B surface antigen (HBsAg) with an HBV DNA copy number greater than the upper limit of normal values in the laboratory department of the study center; or (11) Positive hepatitis C virus (HCV) antibody with an HCV RNA copy number greater than the upper limit of normal values in the laboratory department of the study center; or (12) Positive hepatitis C virus (HCV) antibody with an HCV RNA copy number greater than the upper limit of normal values in the laboratory department of the study center. ⑪Conditions that, in the opinion of the investigator, may affect the safety or compliance with the study drug therapy, including but not limited to large pleural/peritoneal/pericardial effusions, uncorrectable pleural/peritoneal/pericardial effusions, psychiatric disorders, etc. ⑪Known hypersensitivity or delayed hypersensitivity to certain components of the recombinant humanized anti-HER2 monoclonal antibody-MMAE coupling agent vedicizumab (Edisil, RC48) for injection or similar drugs Hypersensitivity or delayed hypersensitivity reactions; ⑬Women who are pregnant or breastfeeding or women/men who are planning to have children

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-06-07 (Estimated); Primary Completion 2025-06-06 (Estimated); Study Completion 2026-06-06 (Estimated)

PRIMARY OUTCOMES:
ORR | 8 weeks
  ORR definition: the proportion of patients with tumor volume reduction to pre-specified values (CR/PR) who can maintain the minimum time requirement

SECONDARY OUTCOMES:
PFS | 2 years
  PFS definition: the time from the start of randomization (or the start of treatment in a single-arm trial) to tumor progression or death from any cause, whichever occurs first;
DFS | 2 years
  disease-free survival (DFS) definition: is the time from the start of randomization (or the start of treatment in a single-arm trial) to disease recurrence or death from any cause (whichever occurs first)
OS | 2 years
  OS defined as means the time from the start of randomization (or the start of treatment in a single-arm trial) to death from any cause
complete resection rate | 2 years
  complete resection rate: lesion R0 resection and no extraperitoneal invasion of lymph nodes, no positive lymph on residual
Rate of facial nerve preservation | 2 years
  Rate of facial nerve preservation: the proportion of patients whose facial nerve was originally judged by the surgeon to require surgical resection and who were able to preserve the facial nerve as a result of neoadjuvant or conversion therapy.

IPD SHARING:
Plan to Share IPD: No